CLINICAL TRIAL: NCT04465435
Title: Sustainable UNiversity Life (SUN): Mental Illness and Pain Conditions Among Students - a Cohort Study to Identify Modifiable Risk and Prognostic Factors
Brief Title: Sustainable UNiversity Life (SUN) Study
Acronym: SUN
Status: Active, not recruiting | Type: Observational
Sponsor: Sophiahemmet University (Other)
Collaborators: Karolinska Institutet (Other); Forte (Industry)
Responsible Party: Sponsor
Other Study IDs: FORTE2018-00402
Record Dates: First submitted 2020-06-17; First posted 2020-07-10 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Issue; Musculoskeletal Pain
Keywords: Cohort study; Depression; Anxiety; Stress; Pain; Lifestyle; Students; Risk Factors; Prognostic factors
MeSH Terms: conditions — Musculoskeletal Pain; Depression; Anxiety Disorders; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SUN-participants: University students enrolled in a selected university in Stockholm, studying on a full-time educational program with at least one academic year left before graduation.
  There is no intervention. The exposures are repeated measures, 5 times (every three months), using web-based self-report questionnaires during one academic year. Also weekley SMS are used to measure depression, anxiety and pain intensity.
  Interventions: Other: Web-based self-report questionnaires; Other: Focus Group Interviews

INTERVENTIONS:
Other: Web-based self-report questionnaires — Web-based self-report questionnaires based on well established instruments.
Other: Focus Group Interviews — Group conversation with open-ended questions with 7-10 students/group on topics relevant to the aim of the study.

SUMMARY:
In 2017, Socialstyrelsen reported that mental ill-health in young adults had increased by almost 70% in the previous10 years. A 2014 report showed that 5% of men and 11% of women 18-24 years were diagnosed with depression or anxiety in Stockholm County. Furthermore, 41% of women 21-24 years have self reported psychological distress. Regarding pain, 28% of men and 36% of women 16-24 years have disabling neck pain. Little is known about the etiology and prognosis of poor mental health in university students.

The aim is to advance knowledge about the etiology of depression, anxiety, stress and pain in undergraduate university students. The investigators will study a cohort of students at full-year programs at universities in the Stockholm area. Primary research questions are whether modifiable factors such as sleep quality, lifestyle, screen time and work environment are independent risk factors for incident episodes or unfavorable trajectories of depression, anxiety and pain in men and women? To be able to answer these research questions we designed a prospective cohort study targeting 5000 university students.

DETAILED DESCRIPTION:
Study objectives:

The overall study aim is to advance the knowledge about the etiology and prognosis of common mental health problems (depression, anxiety and stress) and musculoskeletal pain experienced by undergraduate university students in Sweden.

Specific research questions:

Are modifiable factors as bad sleep quality, meal patterns, low physical activity/sedentary lifestyle, pain conditions and bad study environment independent risk factors of incident episodes of troublesome depressive and anxiety symptomatology and musculoskeletal pain and of unfavorable trajectories of depressive, anxiety, stress and pain symptoms? Are modifiable factors as bad sleep quality, meal patterns, low physical activity/sedentary lifestyle, pain conditions and bad study environment independent prognostic factors for recovery from troublesome depressive and anxiety symptomatology and musculoskeletal pain? Do such potential risk factors and trajectories vary between men and women? What are the trajectories of sleep quality, meal patterns, physical activity/sedentary lifestyle, pain and substance use during one academic year (describe the fluctuations of risk factors)?

Study design:

Cohort study of undergraduate or graduate (up to master level) full time program students, 18 years of age or older, with at least one academic year before graduation, followed-up four times during an academic year.

Source populations:

The source populations for this project are undergraduate or graduate (up to master level) full-time program students, 18 years of age or older, with at least one academic year before graduation at universities in the Stockholm area.

Data collection:

Data collection will be performed with questionnaires through a link sent to students e-mail address, provided by the participating universities. The students will be able to access the questionnaire for a four-week period at baseline and each follow-up.

Exposures:

Sleep quality, physical activity and sedentary behavior, substance use in the past three months (non-medical use), study environment, body image, perfectionism, gambling, compulsive exercise, social media use, cyberbullying, procrastination and loneliness.

Outcomes:

Outcomes will be measured with the Depression Anxiety Stress Scales-21 (DASS-21). The DASS-21 includes three subscales designed to measure depression, anxiety and stress symptoms in non-clinical populations with response alternatives on a Likert scale ranging from 0-3. Higher scores indicate more severe symptoms. Musculoskeletal pain will be measured with the The Nordic Musculoskeletal pain Questionnaire (NMQ) that cover most potential musculoskeletal pain sights. The questionnaire measure musculoskeletal symptoms, and pain intensity in nine body areas: the neck, shoulder, elbow, wrists/hands, upper back, lower back, hips/thighs/buttocks, knees and ankle/feet. The questions were modified to ask about the previous month rather than the previous 12 months as per the original NMQ. Those reporting no symptoms were assigned a pain score of zero, while those who reported having musculoskeletal symptoms were also asked to report how intense pain was on average over the last month, on a scale from zero, which refers to no complaints, to nine, which refers to the pain 'as bad as it can be'.

Potential confounders:

The investigators will collect the following variables as potential confounders of the association between the exposures and the outcomes. These confounders were selected based on our review of the literature.

Sociodemographic variables: age, gender, citizenship, marital status, number of dependents, parents' marital status, parents' employment status, annual personal and household income, hours of work per week, living arrangement, and commute time.

Academic variables: Overall average in the past year (first year students will provide the average for the final year of high school), program of study, year of study.

General health and medically diagnosed comorbidities: The investigators will ask participants to rate their general health and comorbidities diagnosed by a health care provider in the past year. We will selected comorbidities that are reported by > 5% of the sample in our pilot study. In the Canadian pilot study, these include: allergies, arthritis, asthma, attention disorder/learning disability, eating disorder, hypertension, intestinal or stomach ulcers, migraine headaches, mood disorder, scoliosis, and sexually transmitted infections.

Data analysis and statistics:

Definition of trajectories: Trajectories of the outcomes depression, anxiety, stress symptoms and pain will emerge by latent class growth mixture models (LCGMM) that allows for the identification of multiple underlying trajectories within a defined population. In LCGMM, each trajectory is defined by its own growth parameters (intercept, linear slope), which are assumed to be latent. We will use the Baysian Information Criteria (BIC), Bootstrap Likelihood Ratio Test (BLRT) and entropy (measure of uncertainty) to determine whether our 4-trajactory hypothesis offers the best fitting solution for the data. Also trajectories of sleep quality, food insecurity, physical activity/sedentary lifestyle, and substance use will be identified with this method.

Associations between exposures and trajectories: The investigators will use multinomial logistic regression analyses to determine the associations between each of the exposures and trajectories of outcomes. The investigators will report the associations as odds ratios (OR) and 95% confidence intervals (95% CI). The investigators will first build bivariate models to measure the crude associations between the exposures and trajectories. To identify confounders, the investigators will build models to test whether the inclusion of each potential confounder produced a ≥ 10% change in any of the associations.

Associations between exposures and incident cases of depression, anxiety, stress symptoms and pain: At baseline, the investigators will identify a sub-cohort of students at risk of developing troublesome depressive and anxiety symptoms and pain respectively. The investigators will use Kaplan-Meier estimates to describe the incidence and discrete time survival analysis to measure the associations between the exposures and the outcome. In all models, the reference category will be the level of exposure hypothesized to be associated with the lowest risk of the outcome. ORs and 95% CIs will be used to describe the strength and direction of association. The same approach as described above will be used to identify prognostic factors (starting with a sub-cohort under "risk" of recovery) and for control for confounding.

Sample size: The investigators estimated the number of parameters that could be included in the multinomial logistic regression models based on distributions of participants across the four hypothesized trajectories (no symptoms; improvement; worsening; and persistent) using two diverse distribution scenarios. In scenario 1, we hypothesized that 70% have no symptoms, 13% experience worsening, 10% improve and 7% have persistent symptoms. In scenario 2, the investigator hypothesized equal distribution (25%) across trajectories. Based on these assumptions, the investigators estimated that the models could accommodate between 32 parameters if the investigators recruit 1000 students (scenario 1) to as many as 234 parameters if the investigators recruit 5000 participants (scenario 2).

Covid-19 sub-study:

The recruitment and data collection for the cohort study took place before and during the Covid-19 pandemic.Therefore, the investigators started a more fequent recording of levels of pain, axiety and depression from May 2020 with weekly text messages. The data Collection before and during the pandemic provide a chance to investigate the change in symptoms of depression, anxiety and stress and lifestyle behaviors in relation to the pandemic. The specific research questions with regards to this Covid-19-related sub-study are: 1) Are there any changes regarding symptoms of mental health problems during the first month of the pandemic? 2) Will students display changes in healthy lifestyle behaviors such as sleep patterns and quality, meal pattern, exercise and substance use during the first month of the pandemic and 3) Different trajectories of symptoms of low mood, worry and pain during the course of the pandemic will be measured weekly with the aim of identifying factors related to unfavorable trajectories.

ELIGIBILITY:
Inclusion Criteria:

Students at selected universities/colleges in the Stockholm area attending selected educational programs with at least one remaining academic year before graduating. Students from matriculation to master level studies are invited to participate. Participants need to be 18 years of age or older, have access to a smart phone, laptop or tablet and speak sufficient Swedish or English.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — All students invited to participate in the study answer the question about gender identity - female, male or other. All analyses with regard to gender in the study are based on self-representation based on these three categories.
Study Population: University students attending selected universities in Stockholm, Sweden. A number of universities are included representing different educational programs such as medicine and life sciences, business, social sciences and technology. There is a majority of student from medical. and life science educational programs. The aim is to include a total of 5000 students.
Sampling Method: Non-Probability Sample
Enrollment: 4262 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal pain | 2019-2022
  Repeated measures with web-based questionnaires, 5 times (every 3 months), over one year. Outcome measures: Musculoskeletal pain will be measured with the The Nordic Musculoskeletal Questionnaire (NMQ). The NMQ measure musculoskeletal symptoms, and pain intensity in nine body areas: neck, shoulder, elbow, wrists/hands, upper back, lower back, hips/thighs/buttocks, knees, ankle/feet. The questions were modified to assess previous month rather than the previous 12 months as per the original NMQ. No symptoms = a pain score of 0, while the participants who report musculoskeletal symptoms also report average pain intensity over the last month, on a scale from 0 (no complaints), to 9 (pain 'worst possible'). Weekly text messages measure levels of pain.
Mental health problems | 2019-2022
  Repeated measures with web-based questionnaires, 5 times (every 3 months), over one year. Outcome measures: Depression Anxiety Stress Scale-21(DASS-21). DASS-21 includes three subscales (range 0-3, score 0-63, higher scores = more symptoms) to measure depression, anxiety and stress symptoms in nonclinical populations. Weekly text messages measure levels anxiety and depression.

SECONDARY OUTCOMES:
Pain related to the Covid-19 pandemic. | 2019-2020
  Web-based questionnaires comparing students entering the study before the Covid-19 pandemic and after. Outcome measures: Musculoskeletal pain will be measured with the The Nordic Musculoskeletal Questionnaire (NMQ). The NMQ measure musculoskeletal symptoms, and pain intensity in nine body areas: neck, shoulder, elbow, wrists/hands, upper back, lower back, hips/thighs/buttocks, knees, ankle/feet. The questions were modified to assess previous month rather than the previous 12 months as per the original NMQ. No symptoms = a pain score of 0, while the participants who report musculoskeletal symptoms also report average pain intensity over the last month, on a scale from 0 (no complaints), to 9 (pain 'worst possible'). Weekly text messages measure levels of pain.
Mental health problems related to the Covid-19 pandemic. | 2019-2020
  Web-based questionnaires comparing students entering the study before the Covid-19 pandemic and after. Outcome measures: Depression Anxiety Stress Scale-21(DASS-21). DASS-21 (3 subscales, range 0-3, score 0-63, higher scores = more symptoms) to measure depression, anxiety and stress symptoms in nonclinical populations. Weekly text messages measure levels of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Skillgate, Professor, Ph.D., Principal Investigator — Sophiahemmet
Locations (1):
- Sophiahemmet University, Stockholm, SE, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Parallell studies in Norway and Canada have been planned for cross-cultural comparisons with merged data sets.

REFERENCES:
- [Background] Edlund K, Sundberg T, Johansson F, Onell C, Rudman A, Holm LW, Grotle M, Jensen I, Cote P, Skillgate E. Sustainable UNiversity Life (SUN) study: protocol for a prospective cohort study of modifiable risk and prognostic factors for mental health problems and musculoskeletal pain among university students. BMJ Open. 2022 Apr 4;12(4):e056489. doi: 10.1136/bmjopen-2021-056489. PMID 35379630
- [Derived] Larsson K, Onell C, Edlund K, Kallberg H, Holm LW, Sundberg T, Skillgate E. Lifestyle behaviors in Swedish university students before and during the first six months of the COVID-19 pandemic: a cohort study. BMC Public Health. 2022 Jun 16;22(1):1207. doi: 10.1186/s12889-022-13553-7. PMID 35710368
- [Derived] Edlund K, Johansson F, Lindroth R, Bergman L, Sundberg T, Skillgate E. Body image and compulsive exercise: are there associations with depression among university students? Eat Weight Disord. 2022 Oct;27(7):2397-2405. doi: 10.1007/s40519-022-01374-x. Epub 2022 Feb 18. PMID 35179726